CLINICAL TRIAL: NCT03867435
Title: Assessing Clinical Endpoints and Biomarkers in Myotonic Dystrophy Type-1 and Type 2
Brief Title: Assessing Clinical Endpoints and Biomarkers in Myotonic Dystrophy Type-1 and Type 2 (ASCEND-DM)
Status: Terminated | Type: Observational
Why Stopped: PI left the NIH
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190065; 19-N-0065
Record Dates: First submitted 2019-03-02; First posted 2019-03-08 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Myotonic Dystrophy Type-1; Myotonic Dystrophy Type-2
Keywords: Muscle Weakness; Muscular Dystrophy; Neuromuscular Disease; Myotonia
MeSH Terms: conditions — Muscle Weakness; Muscular Dystrophies; Neuromuscular Diseases; Myotonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Individuals with DM1: Individuals with myotonic dystrophy type 1 (DM1)
- Individuals with DM2: Individuals with myotonic dystrophy type 2 (DM2)

SUMMARY:
Background:

Myotonic dystrophy is a long-term genetic disorder that affects muscle function. Symptoms include gradually worsening muscle loss and weakness. Muscles often contract and cannot relax. Researchers want to find out how various tests for DM1 or DM2 change over 2 years, to help them develop better tests for people with these diseases. Data and samples from this study will be shared with the Myotonic Dystrophy Clinical Research Network (DMCRN) investigators participating in the ongoing Establishing Biomarkers and Clinical Endpoints in Myotonic Dystrophy Type 1 (ENDDM1) study

Objective:

To find better ways to assess how myotonic dystrophy type 1 or type 2 affects people.

Eligibility:

People ages 11 70 with DM1 or DM2

Design:

Participants will have 3 study visits over 2 years. Participants may be admitted to the clinic. Each visit may last up to a week and will include:

Medical history and physical exam

Blood, heart, and pregnancy tests

Questions about their disease

Breathing and muscle tests, including tests of movement, grip, and hand opening

Speech and swallowing exam

Magnetic resonance imaging (MRI). Participants will lie on a table that slides into a cylinder.

A magnetic field and radio waves will take pictures of the body. They may do a task during the scan. They may have a dye injected.

Pictures of chemicals in the brain or muscle taken in an MRI scanner

Thinking and memory tests

Sleep studies. Electrodes placed on the scalp will record the electrical activity of the brain.

Other devices on the body will measure heartbeat, breathing, movement, and oxygen.

Tests of electrical activity of muscles. Participants move their arms and legs with disks stuck on their skin.

Visits may also include:

Exam by a physician expert in stomach and bowel disorders

A piece of muscle and/or spinal fluid removed by needle

Sponsoring Institute: National Institute of Neurological Disorders and Stroke

...

DETAILED DESCRIPTION:
Objective: Myotonic dystrophy type 1 (DM1) and type 2 (DM2) are the most common inherited skeletal myopathies in adults. RNA toxicity is the core disease mechanism, good molecular targets have been identified and there has been rapid progress in developing targeted therapies. However, incomplete characterization and limited biologic understanding of phenotypic heterogeneity, and lack of reliable clinical endpoints and biomarkers remain major obstacle in the road to therapeutic success in these diseases. The present study seeks to overcome these roadblocks building on previous work of the Myotonic Dystrophy Clinical Research Network (DMCRN) (14-N-0132 study) with the following added features: 1) larger DM1 cohort including 11 - 70 year old individuals; 2) including DM2 individuals, 3) longer study duration; 4) allowing validation of NIH custombuilt devices for longitudinal measurements; and 5) including non-muscle endpoints and biomarkers specifically respiratory and central nervous system (CNS) function, which are important for survival and quality of life. The goal of the current study is to prospectively assess the disease progression over 2 years in individuals with DM1 and DM2. Selected tests, imaging and patient-reported outcomes will be assessed for ability to quantify disease burden, detect disease progression and predict changes. Additionally, we will examine muscle and cerebrospinal fluid (CSF) RNA alternative splice events as biomarkers of DM1 and DM2 severity and explore genetic modifiers of DM1 and DM2 severity by genome wide association (GWA) study.

Study population: This study plans to enroll up to 180 participants: 120 individuals with DM1 and 60 individuals with DM2 (open to both juvenile and adult individuals (11 to 70 years old, inclusive)) at the NIH Clinical Center.

Study Design: This will be a prospective observational study. No treatment will be administered as part of this study. Participants will receive standard of care as determined by their treating physician. Participants will report to the NIH Clinical Center for 3 visits each: at baseline (Visit 1), at 1-year from baseline (Visit 2), and at 2-years from baseline (Visit 3). To reduce fatigue and impact on results, each study visit be split into more than one trip to the NIH within a 30 day window) and may require the patient to be admitted to the clinical center. Each trip to the NIH for a study visit may last up to seven days. Study procedures for each visit are outlined in Section 4 and Appendix A. Data and samples will be shared with DMCRN investigators participating in Establishing Biomarkers and Clinical Endpoints in Myotonic Dystrophy Type 1 (ENDDM1) study as indicated in Appendix B.

Outcome measures: No specific primary and secondary outcomes will be specified; however, the change in the following measures from baseline may be used to characterize the baseline status and disease progression over the course of the study: 1) muscle strength; 2) myotonia; 3) hand and upper arm functional tests; 4) measures of gait, balance and mobility; 5) skeletal muscle MRI measures of muscle mass and fatty degeneration; 6) skeletal muscle RNA biomarkers from biopsied tissue; 7) cognitive function; 8) brain MRI measures of gray matter volume, white matter hyperintensity volume, whole brain volume, integrity of white matter tracts measured as mean diffusivity and fractional anisotropy and resting state functional connectivity by functional MRI; 9) pulmonary function tests; 10) MRI measures of the diaphragm motion and contractility, myocardial function as well as myocardial fat and water composition and fibrosis; 11) clinical assessments of sleep, speech and swallow and gastrointestinal motility impairment; and 12) CSF RNA biomarkers and genetic modifiers of DM1 and DM2 severity from a GWA study in collaboration with other DMCRN researchers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 11 to 70 inclusive
* Competent to provide informed consent and assent (consent of a parent or guardian will be required for pediatric participants)
* Positive genetic test for DM1 or DM2 (Genetic testing for DM1 or DM2 may be determined after enrollment

EXCLUSION CRITERIA:

* Concurrent enrollment in a clinical trial or participation in an investigative drug trial within 6 months of study entry.
* Concurrent pregnancy or planned pregnancy during the course of the study.
* Concurrent medical condition that would, in the opinion of the investigator or clinical evaluator, compromise performance on study measures:
* Clinically significant infections or medical illness within 30 days from study entry.
* History of, or abnormal laboratory values indicative of, significant medical, neurologic (other than DM1 or DM2), or psychiatric disorders.
* A recent history (30 days prior to study entry) of any of the following conditions on routine blood screening: white blood cells < 3000, platelets < 100,000, hematocrit < 30%, symptomatic liver disease with serum albumin < 3 g/L, or creatinine > 1.5 mg%.
* Any of the following medical conditions: uncontrolled or insulin-dependent diabetes mellitus, congestive heart failure, symptomatic cardiomyopathy, symptomatic coronary artery disease, cancer (other than skin cancer) within 5 years from study entry, multiple sclerosis, or other serious medical illness.
* Other diseases that mimic the signs or symptoms of DM1 or DM2. Coexistence of other neuromuscular disease.
* Thyroid dysfunction that is untreated (if on thyroid hormone replacement therapy, need to have adequate and stable replacement over the previous 6 months from study entry).
* Second or third degree heart block, atrial flutter, atrial fibrillation, ventricular tachycardia, or is receiving medication for the treatment of cardiac arrhythmia.
* Liver or kidney disease requiring ongoing treatment.
* Have a seizure disorder.
* Drug or alcohol abuse within 3 months of study entry (DSM-V criteria will be used for the diagnosis and level of a substance use disorder:
* Treatment with supplemental anabolic hormones (including testosterone, human recombinant growth hormone, human recombinant insulin like growth factor-1, other anabolic drug mixtures) during the previous 12 months from study entry.

Note: non-ambulatory participants are not excluded but are limited to <15% of enrollment. Individuals using a cane or walker will not be examined for gait, balance and mobility.

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
to characterize baseline status and disease progression over two years in the handgrip strength by dynamometry of DM1 and DM2 patients. | one-year and two-years
  strength of handgrip by hand-held force transducer

SECONDARY OUTCOMES:
muscle strength, myotonia, physical function of limbs, MRI changes of muscle fat %, cognition, brain MRI changes, diaphragm function, muscle RNA biomarkers, sleep, speech, swallow, bowel function | one and two years
  changes in the outcome measures described from baseline
CSF RNA biomarkers, genetic modifiers of disease severity | one and two years
  RNA splicing changes using RNA-seq in CSF and Genome-wide association study for genetic variants predicting disease severity in collaboration with DMCRN

CONTACTS AND LOCATIONS:
Overall Officials: Ami K Mankodi, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-N-0065.html